CLINICAL TRIAL: NCT04082858
Title: Ketamine Interleaved With Electroconvulsive Therapy for Depression, A Pragmatic Randomised Controlled Pilot Trial
Brief Title: Ketamine Interleaved With Electroconvulsive Therapy for Depression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate recruitment due to COVID-19
Sponsor: St Patrick's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Prof Declan McLoughlin, Professor, St Patrick's Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 11/18
Record Dates: First submitted 2019-08-19; First posted 2019-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Depression
Keywords: Ketamine; Electroconvulsive Therapy; Depression; ECT
MeSH Terms: conditions — Depression | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Pragmatic, randomised, controlled, parallel group, pilot clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants will receive twice-weekly infusions of ketamine at 0.05mg/kg for the duration of treatment with ECT. All infusions will be administered by a Consultant Anaesthetist.
  Interventions: Drug: Ketamine
- Midazolam (Active Comparator): Participants will receive twice-weekly infusions of midazolam at 0.045mg/kg for the duration of treatment with ECT. All infusions will be administered by a Consultant Anaesthetist.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine — A sub-anaesthetic dose of ketamine will be administered in twice-weekly infusions
  Other Names: Ketalar
  Arms: Ketamine
Drug: Midazolam — A sub-anaesthetic dose of midazolam will be administered in twice-weekly infusions
  Other Names: Hyponovel
  Arms: Midazolam

SUMMARY:
Pragmatic, randomised, controlled, parallel group, pilot clinical trial of ketamine vs. midazolam interleaved with electroconvulsive therapy (ECT) as an adjunctive treatment for a major depressive episode. The main purpose of the pilot study is to assess trial processes to help inform a future definitive trial.

DETAILED DESCRIPTION:
Patients referred for treatment with ECT at St Patrick's Mental Health Services for treatment of a depressive episode will be eligible for recruitment to the clinical trial. Participants will be invited to be randomised to a course of twice-weekly ketamine or midazolam infusions for the duration of ECT. Participants will receive the first allocated infusion following the first or second treatment with ECT. Block randomisation will be independently performed. Infusions will be delivered on separate days to ECT. Physical, psychotomimetic and cognitive outcomes will be monitored before, during and after infusions.Treatment-as-usual will continue throughout the entire trial.

Trial Interventions: participants will receive twice-weekly infusions of either ketamine at 0.5mg/Kg or midazolam at 0.045mg/Kg. All infusions will be administered by a Consultant Anaesthetist. Repeated infusions of allocated drug have been shown to be safe and well tolerated by patients with mental illness. Minor haemodynamic changes and psychotomimetic side effects can occur and will be assessed regularly during infusions and for 120 minutes afterwards. Participants will be followed-up at six weeks and three months after the final infusion to assess for relapse according to standardised criteria.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Able to provide informed consent
* Voluntary admission for treatment of an acute depressive episode
* Meet DSM-V criteria for a major depressive disorder (MDD) and bipolar affective disorder (current episode depression)
* Montgomery Asberg Depression Rating Scale 10 item version (MADRS) score of ≥20
* Referred for treatment with ECT
* Sufficiently physically healthy to receive ketamine/midazolam and ECT

Exclusion Criteria:

* Inability to provide informed consent
* Current involuntary admission
* History of Axis 1 diagnosis other than major depression
* Medical condition rendering unfit for ECT
* Active suicidal intention
* Presence of major neurological or organic brain disorder
* Alcohol/substance dependence in previous six-months
* Pregnancy or inability to confirm use of adequate contraception during the trial
* Breastfeeding women
* Contraindications to ketamine
* Contraindications to midazolam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 18 weeks
  A validated, 10-item, depression rating scale to measure depressive symptomatology and response to treatment. During the infusion sessions MADRS scores will be obtained immediately pre-infusion and at +60 and +120 minutes afterwards. Depression measures will be repeated at week 6 and at three-months post infusion. This outcome measure assesses the change in MADRS scores during the pilot trial.
  A course of ECT can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. Participants will be followed up for three months (12 weeks) after their final infusion. In total, participants outcome measures will be repeated for up to 18 weeks.

SECONDARY OUTCOMES:
The Quick Inventory of Depressive Symptoms, self-report version (QIDS-SR16) | 18 weeks
  The QIDS-SR16 is a validated self-report measure of depressive symptoms. This consists of 16 questions rated 0-3. Its score range is 0-48, with higher scores reflecting greater burden of depressive symptoms.
  During the infusion sessions in the pilot trial QIDS scores will be obtained immediately pre-infusion and at +60 and +120 minutes afterwards. For longer-term follow-up, depression measures will be repeated at weeks 6 and three-month follow-up.
  A course of Electroconvulsive Therapy (ECT) can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. Participants will be followed up for three months (12 weeks) after their final infusion. In total, participants outcome measures will be repeated for up to 18 weeks (12 weeks + 6 weeks).
The Clinician-Administered Dissociative States Scale (CADSS) | 6 weeks
  The CADSS measures dissociative symptoms. It will be administered before, during and after infusions in order to capture the range of possible subjective side effects of either agent. This consists of 23 questions and scores for each question range from 0-4. The maximum score is 92 with higher scores indicating more dissociative symptoms.
  Participants will have the CADSS performed before, during (+30mins) and after (+60mins) each infusions.
  A course of Electroconvulsive Therapy (ECT) can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. The above measures will be repeated for the duration of the trial i.e. for up to 6 weeks.
The Brief Psychiatric Rating Scale (BPRS) | 6 weeks
  The BPRS measures psychotomimetic effects. The investigators will use the positive symptoms subscale of the Brief Psychiatric Rating Scale. The 4-item positive symptoms subscale measures suspiciousness, hallucinations, unusual thought content, and conceptual disorganisation. Each question is scored between 0-7. The maximum score in this 4-item questionnaire is 28. Higher scores indicate more severe psychotic symptoms.
  Participants will have the BPRS performed before, during (+30mins) and after (+60mins) each infusion.
  A course of Electroconvulsive Therapy (ECT) can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. The above measures will be repeated for the duration of the trial i.e. for up to 6 weeks
Young Mania Rating Scale (YMRS; mood item) | 6 weeks
  Investigators will use the mood item of them YMRS to assess for psychotomimetic effects. This item is rated 0-4. The higher scores reflect elevated mood.
  Participants will have the YMRS performed before, during (+30mins) and after (+60mins) each infusion.
  A course of Electroconvulsive Therapy (ECT) can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. The above measures will be repeated for the duration of the trial i.e. for up to 6 weeks
The Patient-Rated Inventory of Side Effects (PRISE) | 6 weeks
  The PRISE will be used to document other general adverse events by patients before, during and after infusions. This is a patient self-report used to qualify side effects by identifying and evaluating the tolerability of each symptom. It is a 9 item assessment.
  Participants will have the PRISE performed before, during (+30mins) and after (+60mins) each infusion.
  A course of ECT can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. The above measures will be repeated for the duration of the trial i.e. for up to 6 weeks
The Montreal Cognitive Assessment (MoCA) | 18 weeks
  The MOCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, conceptual thinking, calculations, and orientation. It is scored out of a maximum of 30. The higher scores indicate better cognition.
  The MOCA will be performed at baseline, one day after the first and final infusions and at 12 weeks after the final infusion.
  A course of Electroconvulsive Therapy (ECT) can be prescribed for a maximum to 6 weeks (12 sessions in total, twice weekly for 6 weeks). Trial infusions will be administered twice weekly on separate days to ECT, for the duration of treatment with ECT. Therefore, trial infusions may be administered for up to 6 weeks. Participants will be followed up for three months (12 weeks) after their final infusion. In total, participants outcome measures will be repeated for up to 18 weeks (12 weeks + 6 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Declan McLoughlin, PhD, Principal Investigator — St Patrick's Hospital
Locations (1):
- St Patrick's University Hospital, Dublin, Co. Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No